CLINICAL TRIAL: NCT01833923
Title: A Phase I Study of Anlotinib on Tolerance and Pharmacokinetics
Acronym: ALTN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Collaborators: Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-I-01
Record Dates: First submitted 2013-03-29; First posted 2013-04-17 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Advanced Cancer
Keywords: Advanced cancer
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anlotinib (Experimental): dosage form:capsule dosage:5mg,10mg,16mg,12mg frequency:once one day duration:Continuous two weeks then stop a week
  Interventions: Drug: anlotinib

INTERVENTIONS:
Drug: anlotinib — oral medicine.
  Other Names: ALTN

SUMMARY:
Anlotibib (ALTN) is a kind of innovative medicines approved by State Food and Drug Administration（SFDA） which was researched by Jiangsu Chia-tai Tianqing Pharmaceutical Co., Ltd.

ALTN is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR2 and VEGFR3. It has the obvious resistance to new angiogenesis.

DETAILED DESCRIPTION:
The primary objective of this trial is to explore the maximum tolerated dose(MTD), dose-limiting toxicity(DLT) of ALTN and rational dosage regimen for phase II study, to investigate the pharmacokinetics with single and multiple doses of ALTN from 5mg/d,10mg/d,16mg/d,12mg.

ELIGIBILITY:
Inclusion Criteria:

1. late malignant tumor patients diagnosed with the pathological and/or cytological;
2. lack of the standard treatment or treatment failure;
3. 18-65years, ECOG:0-1,Expected survival period >3 months;
4. stop medicine > 30 days if any other chemotherapy drugs be used.
5. HB≥90g/L,ANC(Absolute Neutrophil Count) ≥1.5×109/L；PLT ≥100×109/L ,BIL/ALT/AST(aspartate aminotransferase )/Cr in normal range,or CCR≥60ml/min,TG≤ 3.0mmol/L，cholesterol≤7.75mmol/L; LVEF≥LLN.
6. Female should be agreed to use contraceptive during the study and after 6 months (such as intrauterine device(IUD), the pill or a condom); The serum or urine pregnancy test negative before take ALTN, and is out of non-lactation period. Male should be agreed to use contraceptive during the study and after the period of 6 months.
7. Volunteer, informed consent form (ICF) signed, compliance.

Exclusion Criteria:

1. Subject was diagnosed with other malignant tumors previously or meanwhile;
2. Participated in other clinical trials in four weeks;
3. Has influence of oral drugs(such as unable to swallow, gastrointestinal tract after resection);
4. Already diagnosed with brain metastases, spinal cord compression, cancerous meningitis, or screening CT or MRI findings of the brain or soft meningeal disease patient;
5. Hypertension
6. Urine protein: ++, and urinary in 24 hours > 1.0g;
7. Coagulant function abnormality: subject with bleeding tendency (such as active peptic ulcer) or are receiving thrombolysis or anticoagulant therapy;
8. Subject with psychiatric drugs abuse history and can't get rid of, or mental disorder;
9. With artery/venous thrombotic before oral ALTN;
10. With history of anticoagulant, vitamin K antagonists(such as warfarin or heparin) or other analogues treatment;
11. With Abnormal thyroid function;
12. With history of psychiatric drugs abuse or a mental disorder;
13. Viral hepatitis B or hepatitis c patients (including hepatitis b, hepatitis c virus carriers);
14. Have immunodeficiency history;
15. According to the researcher's judgment,there are concomitant diseases which will seriously endanger the patients or obstruct the patients to complete the clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Tmax Cmax t1/2 AUC | Up to 52 days
  To collect point with single drug:H0/H0.5/H1/H2/H4/H8/H12/H24/H48/H72/H96/H120/H144/H/H168/H192/H216/H240
  To collect point with multiple drug:d1/d2/d4/d7/d10/d14/d15/d21/d22/d28/d35/d42

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 21 days
  blood examination, urine examination, stool examination, blood biochemical (ALT, AST, TB(total bilirubin), DB, BUN, Cr, blood electrolyte), electrocardiogram (ecg), thyroid function, the function of blood coagulation, etc

OTHER OUTCOMES:
tumor size | Up to 42 days
  To evaluate the effectiveness of ALTN by enhanced CT scan every two cycles. Refer to recist 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Yihebali Chi, doctor, Principal Investigator — Cancer Institude and hospital,CAMS
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China